CLINICAL TRIAL: NCT05131620
Title: Virtual Reality and Acupressure Applications in the Catheter Extraction Process in Patients Undergoing Coronary Angiography; Effect on Pain, Anxiety, Vital Signs and Comfort
Brief Title: Virtual Reality and Acupressure Applications; Effect on Pain, Anxiety, Vital Signs and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Esma Gökçe, Principal Investigator (MSc), Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0000-0001-9581-6958
Record Dates: First submitted 2021-09-25; First posted 2021-11-23 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Pain; Anxiety; Vital Signs; Virtual Reality
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: 3 Group randomized
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Venture in the Virtual Reality Group (Experimental): Informed consent form will be signed by the patients who will be included in this group as a result of randomization, and a personal information form and STAI will be filled. After CAG, 10 minutes before the catheter extraction, the patients will be selected from videos such as park and nature walks, beach and seaside walks, underwater, museum tour, and virtual reality glasses will be put on and will be worn during the procedure. In the literature, VR glasses were put on 5-10 minutes before the procedure, continued throughout the procedure, and used for a total of 30-60 minutes. Catheter extraction takes approximately 15-20 minutes and it is planned to continue the virtual reality glasses viewing period for 30 minutes. VAS will be applied during the catheter extraction process, and VAS, SAI and PCS will be applied to all patients after catheter extraction. Vital signs of patients will be recorded before, during and after catheter extraction.
  Interventions: Procedure: Virtual Reality
- Venture in the Acupressure Group (Experimental): Initiative in the Acupressure Group Informed consent form will be signed by the patients who will be included in this group as a result of randomization, and a personal information form and STAI will be filled. Acupressure will be applied 10 minutes before catheter extraction after CAG. Catheter extraction takes approximately 15-20 minutes. VAS will be applied during the catheter extraction process, and then VAS, SAI and PCS will be applied to all patients. Vital signs of patients will be recorded before, during and after catheter extraction.
  Interventions: Procedure: Acupressure
- Control Group (No Intervention): Informed consent form will be signed by the patients who will be included in this group as a result of randomization, and a personal information form and STAI will be filled. Routine application will be made. VAS will be applied during the catheter extraction process, and then VAS, SAI and PCS will be applied to all patients. Vital signs of patients will be recorded before, during and after catheter extraction.

INTERVENTIONS:
Procedure: Virtual Reality — It is planned that VR glasses are put on 5-10 minutes before the procedure and continued throughout the procedure, and the total monitoring time will continue for 30 minutes.
  Arms: Venture in the Virtual Reality Group
Procedure: Acupressure — Acupressure will be applied 10 minutes before catheter extraction after CAG.
  Arms: Venture in the Acupressure Group

SUMMARY:
Coronary angiography (CAG) is an invasive method for imaging the coronary arteries. The femoral artery is frequently used during CAG and patients feel pain and anxiety during removal of the catheters placed in the femoral region. These disorders also negatively affect the vital signs and comfort levels of patients.

Different methods are used in direct proportion to the development of technology for relieving anxiety and pain caused by invasive surgical procedures in patients. These methods include virtual reality (VR) applications. Innovative, up-to-date and original, virtual reality is the fusion of fiction and technology with reality and imagination. These programs; It is stated that in addition to reducing the patient's anxiety and pain, it makes them feel safe, increases their comfort, care satisfaction and positively affects their participation in care.

Acupressure is one of the most widely used non-pharmacological methods to reduce pain and anxiety, and one of the applications included in the Nursing Interventions Classification (NIC). Applications made with manipulations such as pressure and rubbing on certain points on the meridians where energy flow takes place in the body are called acupressure. It has been determined that acupressure applications in different areas reduce pain and anxiety and positively affect vital signs and patient comfort.

Although there are studies in the literature in which different non-pharmacological methods are applied to reduce pain and anxiety caused by catheter extraction after CAG, positively affect vital signs, and increase the level of comfort, no research has been found in which acupressure method and virtual reality methods developed with today's technology are applied together. In this study, it was planned to reduce the pain and anxiety of the patients, to observe the effects on vital signs, and to increase their comfort levels, with acupressure application and virtual reality methods, which have not been applied non-pharmacologically until now, in patients who underwent CAG.

DETAILED DESCRIPTION:
Before starting the research, permission was obtained from Çukurova University Medical Faculty Balcalı Hospital Cardiology Departmant, from Balcalı Hospital Chief Physician, and Çukurova Ethics Committee by the investigator . University Faculty of Medicine Non-Interventional Research Ethics Committee approval was received with the date and number of 02.10.2020/104 An application was made to the Scientific Research Projects Unit to support the project with all permissions. It has been approved as a Scientific Research Project.

Type of Research:

The study was planned as an experimental, randomized controlled trial with 3 groups.

Place and Date of the Research:

The study will be applied to patients who underwent coronary angiography in the Cardiology Department of Çukurova University Medical Faculty Balcalı Hospital October 2021. Cardiology department consists of 1 outpatient clinic, 1 intensive care unit, 1 service, 2 angiography laboratories and 46 patient beds.

Universe and Sample:

The universe of the research will be all patients who will undergo CAG in the Cardiology Department of a university hospital date 2021. A pilot study will be conducted for sampling purposes and 9 patients from each group will be recruited and completed with a total of 27 patients. Patients will be divided into 3 groups (2 experiments, 1 control) by computer randomization.

Data Collection Tools In the collection of data, Informed Voluntary Consent Form (IVCF), Personal Information Form (PIF), Visual Assessment Scale for pain (VAS-Visuel Analog Scale), State-Trait Anxiety Inventory for anxiety (STAI) was created by the researcher by scanning the literature. Perianesthesia Comfort Scale (PCS) will be used for comfort and vital signs will be measured.

Statistical analysis of the collected data will be done using a package program called SPSS (IBM SPSS Statistics 24).

ELIGIBILITY:
Inclusion Criteria:

* Accepting the research
* Able to communicate in Turkish
* Patients whose clinical condition is stable
* between 18 and 88 years old
* No hearing problem
* CAG applied for the first time
* Undergoing a femoral intervention by placing a catheter in their femoral regions
* Those who have no previous psychiatric or mental illness

Exclusion Criteria:

* Refusal to participate in the research
* Complication developed during the operation

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Nonpharmacological method effects (pain) | [Time Frame: Primary VAS pain measurement will be taken at approximately 20th minutes, during the ongoing catheter withdrawal phase.]
  In this study, pain levels of all groups will be measured during the catheter extraction procedure and after the end of the catheter extraction procedure in patients undergoing CAG. VAS-Visual Analog Scale was used to measure pain.
  It is a scale that is evaluated by the patients by making markings on a 10 cm or 100 mm horizontal or vertical line (or horizontal line with numbers from 1 to 10), with one end indicating that the patient is very good the other end is very bad.
  In this method, it is explained to the person that there are two end points indicating whether there is pain and that he should mark any point between these points.
  Pain measurement with the first VAS will be done at the time of catheter extraction.
  Yes Pain - No Pain
  1 2 3 4 5 6 7 8 9 10 Figure 1. VAS
Nonpharmacological method effects (Anxiety) | [Time Frame: Primary STAI measurement will be performed before all groups are processed and catheter withdrawal begins. STAI measurement will be at take 0th minute.]
  In this study, the effects on anxiety during catheter extraction in patients undergoing CAG will be measured. Anxiety measurement will be made with STAI (State Trait Anxiety Inventory). The STAI will be filled prior to catheter removal and the state anxiety inventory (SAI) will be refilled after the procedure.
  The scale will be used to evaluate the anxiety levels of patients before and after the procedure. It is intended to describe the state of continuous anxiety and the level of anxiety felt by the individual against the situation he is in. In the scale used, there are 40 items in total, with 20 items examining the individual's state anxiety and 20 items examining trait anxiety. The result of the scale is evaluated as mild anxiety at 20-39 points, moderate anxiety at 40-59 points, severe anxiety at 60-79 points, and panic at 80 points.
Nonpharmacological method effects (Comfort) | [Time Frame: Perianesthesia Comfort Scale (PCS) will be applied after the catheter withdrawal process is completed. PCS measurement will be take at approximately 40th minute.]
  In this study, comfort levels will be measured in patients undergoing CAG after the end of the catheter extraction process in all groups. The Perianesthesia Comfort Scale (PCS) was used to measure comfort.
  It is used to evaluate the expected comfort change state by determining comfort requirements. The scale consists of 24 items that question the self-concept and emotions that reflect the general thought process of the individual regarding the invasive procedure. Each statement in the scale has a Likert-type scoring system ranging from 1 to 6, ranging from "strongly disagree" to "strongly agree". The lowest total score that can be obtained from the scale is 24, and the highest total score is 144.
Nonpharmacological method effects (Vital signs-Systolic and diastolic blood pressure mmHg) | [Time Frame: Systolic and diastolic blood pressures, which are vital signs of the patients, will be recorded at the 0th minute before the catheter extraction, at the 20th minute during and 40th minute afterward.]
  In this study, patients in all groups undergoing CAG; systolic and diastolic blood pressures will be measured before the catheter extraction process begins, while the catheter extraction process is in progress, and after the catheter extraction process is completed.
Nonpharmacological method effects (Vital signs-Respiratory rate per minute) | [Time Frame: Respiratory rate per minute, which are vital signs of the patients, will be recorded at the 0th minute before the catheter extraction, at the 20th minute during and 40th minute afterward.]
  In this study, patients in all groups undergoing CAG; respiratory rate per minute will be measured before the catheter extraction process begins, while the catheter extraction process is in progress, and after the catheter extraction process is completed.
Nonpharmacological method effects (Vital signs-Heart rate per minute) | [Time Frame: Heart rate per minute, which are vital signs of the patients, will be recorded at the 0th minute before the catheter extraction, at the 20th minute during and 40th minute afterward.]
  In this study, patients in all groups undergoing CAG; heart rate per minute will be measured before the catheter extraction process begins, while the catheter extraction process is in progress, and after the catheter extraction process is completed.

SECONDARY OUTCOMES:
Nonpharmacological method effects (pain) | [Time Frame: Secondary VAS pain measurement will be performed at approximately 40th minutes after catheter removal.
  In this study, pain levels of all groups will be measured during the catheter extraction procedure and after the end of the catheter extraction procedure in patients undergoing CAG. VAS-Visual Analog Scale was used to measure pain.
  It is a scale that is evaluated by the patients by making markings on a 10 cm or 100 mm horizontal or vertical line (or horizontal line with numbers from 1 to 10), with one end indicating that the patient is very good the other end is very bad.
  In this method, it is explained to the person that there are two end points indicating whether there is pain and that he should mark any point between these points.
  Pain measurement with the second VAS will be done after the catheter extraction is completed.
  Yes Pain - No Pain
  1 2 3 4 5 6 7 8 9 10 Figure 1. VAS
Nonpharmacological method effects (Anxiety) | Time Frame: The secondary SAI measurement will be made approximately 40th minutes after the catheter withdrawal process of all groups is completed.
  In this study, the effects on anxiety during catheter extraction in patients undergoing CAG will be measured. Anxiety measurement will be made with STAI (State Trait Anxiety Inventory). The STAI will be filled prior to catheter removal and the state anxiety inventory (SAI) will be refilled after the procedure.
  The scale will be used to evaluate the anxiety levels of patients before and after the procedure. It is intended to describe the state of continuous anxiety and the level of anxiety felt by the individual against the situation he is in. In the scale used, there are 40 items in total, with 20 items examining the individual's state anxiety and 20 items examining trait anxiety. The result of the scale is evaluated as mild anxiety at 20-39 points, moderate anxiety at 40-59 points, severe anxiety at 60-79 points, and panic at 80 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Sarıçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No